CLINICAL TRIAL: NCT02227810
Title: Effects of Muscular Electrical Stimulation on Skeletal and Lung Mechanics in Patients With Prolonged Mechanical Ventilation
Brief Title: Electrical Stimulation in Patients With Prolonged Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 103-1702C
Record Dates: First submitted 2014-08-06; First posted 2014-08-28 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2016-03

CONDITIONS: Respiratory Failure
Keywords: Prolong mechanical ventilator,; Electrical stimulation,; Activities of daily life,; Hospitalization outcomes.
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- electrical stimulation (Experimental): Participants will receive muscular electrical stimulation on quadriceps muscle for 20 min/session, twice daily for 10 days
  Interventions: Other: electrical stimulation (high frequency); Other: electrical stimulation (low frequency)
- sham group (Sham Comparator): Participants will receive similar electrical stimulation (ES) procedure as those in intervention group but with ES machine power off.
  Interventions: Other: sham group

INTERVENTIONS:
Other: electrical stimulation (high frequency) — Participants will receive muscular electrical stimulation (75Hz) on quadriceps muscle for 20 min/session, twice daily for 10 days
  Arms: electrical stimulation
Other: electrical stimulation (low frequency) — Participants will receive muscular electrical stimulation (35Hz) on quadriceps muscle for 20 min/session, twice daily for 10 days.
  Arms: electrical stimulation
Other: sham group — Participants will receive similar electrical stimulation (ES) procedure as those in intervention group but with ES machine power off.
  Arms: sham group

SUMMARY:
Muscle atrophy and diaphragm dysfunction are common complication in patients with prolong mechanical ventilator (PMV) and is associated with increased rate of weaning failure and days of hospitalization. Electrical stimulation (ES) has been shown to be beneficial in patients with severe chronic heart failure and chronic obstructive pulmonary disease. The purpose of this study is to examine the effects of ES on skeletal muscle function, pulmonary mechanics and hospitalization outcomes in patients with PMV.

DETAILED DESCRIPTION:
BACKGROUND AND PURPOSE: Muscle atrophy and diaphragm dysfunction are common complication in patients with prolong mechanical ventilator (PMV) and is associated with increased rate of weaning failure and days of hospitalization. Electrical stimulation (ES) has been shown to be beneficial in patients with severe chronic heart failure and chronic obstructive pulmonary disease. The purpose of this study is to examine the effects of ES on skeletal muscle function, pulmonary mechanics and hospitalization outcomes in patients with PMV.

METHODS: Patients who have been on mechanical ventilator for more than 21 days will be recruited from respiratory care center (RCC). All subjects will be randomly assigned into three groups: ES in abdominal muscles (ES-Abd, n=30),ES in brachial biceps (ES-bicep, n=30) and sham group(Sham). Subjects in both groups will receive ES in muscles for 30 min/session, 2 sessions/day for 10 days with the same setting except area of ES. The muscle function will be assessed by skin-fold thickness and muscle strength. The pulmonary function will be assessed by: lung compliance, airway resistance, tidal volume, minute volume and maximal inspiratory pressure. The hospitalization outcome will be followed up until patients are discharged from RCC. The outcomes variables include: weaning rate and duration, mortality, days of ventilator, and length of RCC stay.

ELIGIBILITY:
Inclusion Criteria:

* age>20 years old
* mechanical ventilation for more than 6 h/ day for more than 21 days -- medical stability (arterial blood gas value hydrogen power(pH): 7.35-7.45, atrial oxygen pressure(PaO2): 60 mmHg at 40% fraction of inspired oxygen inspired oxygen fraction (FiO2), absence of signs and symptoms of infection, and hemodynamic stability);

Exclusion Criteria:

* signs of acute infection (BT>38.5℃，WBC>12000 or <3000 per unit
* neuromuscular disease at acute stage
* diagnosis of cancer at end-stage
* pregnancy
* BMI>35kg/m2

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Chi Huang, Principal Investigator — Division of Pulmonary and Critical Care Medicine, Chang Gung Memorial Hospital,Linkou, Taiwan
Locations (1):
- Chang Gung Memorial Hospital, Linkou, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen YH, Hsiao HF, Li LF, Chen NH, Huang CC. Effects of Electrical Muscle Stimulation in Subjects Undergoing Prolonged Mechanical Ventilation. Respir Care. 2019 Mar;64(3):262-271. doi: 10.4187/respcare.05921. Epub 2019 Feb 5. PMID 30723168

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 2012/08/01--2014/07/31 Location: respiratory care center
Period: Overall Study
Arm/Group | Sham Group | Electrical Stimulation
Started | 19 | 34
Completed | 17 | 29
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electrical Stimulation | Sham Group | Total
Number analyzed (Participants) | 34 | 19 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 29 | 13 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.2 (15.4) | 71.9 (17.8) | 74.5 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 20 | 10 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 34 | 19 | 53
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 34 | 19 | 53

OUTCOME MEASURES:

1. Primary Outcome: Level of Activity of Daily Life
Description: The level of activity of daily life was measured by Functional Independence Measure (FIM) score. Possible scores range from 18 (total assist) to 126 (complete independence).
Time Frame: end of intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Group | Electrical Stimulation
Number analyzed (Participants) | 19 | 34
units on a scale | 25.2 (14.5) | 32.0 (21.4)
Statistical Analysis 1: Comparison: Sham Group; Test type: Other; p = 0.652, t-test, 2 sided
Statistical Analysis 2: Comparison: Electrical Stimulation; Test type: Superiority; p = 0.123, t-test, 2 sided

2. Primary Outcome: Muscle Strength
Description: The muscle strength of quadriceps were assessed by Medical Research Council (MRC) scoring system. The MRC score ranges from a 0 points (zero strength) to 5 points (good). The higher points indicated the better muscle strength.
Time Frame: end of intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Group | Electrical Stimulation
Number analyzed (Participants) | 19 | 34
units on a scale | 1.7 (1.1) | 2.7 (1.6)
Statistical Analysis 1: Comparison: Sham Group vs Electrical Stimulation; Test type: Superiority; p = 0.051, t-test, 2 sided
Statistical Analysis 2: Comparison: Electrical Stimulation; Test type: Superiority; p < 0.05, t-test, 2 sided

3. Primary Outcome: Pulmonary Function
Description: The pulmonary function as assessed by the measurement of tidal volume.
Time Frame: end of intervention
Population: t -test
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Sham Group | Electrical Stimulation
Number analyzed (Participants) | 19 | 34
ml | 164.7 (102.7) | 214.4 (57.3)
Statistical Analysis 1: Comparison: Sham Group vs Electrical Stimulation; Test type: Superiority or Other; p = 0.051, t-test, 2 sided

4. Secondary Outcome: Hospitalization Outcomes
Description: The total days that participants stay in the respiratory care center (RCC).
Time Frame: the day participants were discharged from RCC
Population: t test
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sham Group | Electrical Stimulation
Number analyzed (Participants) | 19 | 34
days | 34.2 (18.2) | 32.3 (22.2)
Statistical Analysis 1: Comparison: Sham Group vs Electrical Stimulation; Test type: Superiority or Other; p = 0.792, t-test, 2 sided

ADVERSE EVENTS:
Description: Adverse Events were no collected /assessed.
Arm/Group | Sham Group | Electrical Stimulation
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No